CLINICAL TRIAL: NCT05473936
Title: A Community Health Worker Intervention to Identify and Decrease Barriers to Pre-Procedural COVID 19 Testing Among Los Angeles County Department of Health Safety-Net Patients
Brief Title: A CHW Intervention to Identify and Decrease Barriers to COVID 19 Testing & Vaccination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government); National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1838914-5; 3R01LM012309-04S2 (NIH)
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Vaccine Hesitancy; COVID-19 Testing; Community Health Workers
Keywords: COVID-19 vaccine hesitancy; COVID-19 testing; Community Health Workers; Safety-Net Patients
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm - Standard Treatment (Group 1) (No Intervention): The standard care for the control arm will be: the LACDHS Vaccine Hesitancy Outreach Group calling patients once every month to remind patients of the need to be vaccinated and tested if needed. During the duration of the six weeks, the study participants will be exposed to the call from the LACDHS Vaccine Hesitancy Outreach Group.
  Participants will receive two phone calls six-weeks apart, where they will complete a pre-survey in the first phone call, and 2 surveys (post-survey and CDE survey) in the second phone call. The survey will measure their trust in medical institutions, rate their self-efficacy, and intention, knowledge, and perceptions on COVID-19 testing and vaccination.
- Intervention Arm - CHW-led curriculum (Group 2) (Experimental): Participants assigned to the intervention group will complete the same activities as Group 1 and be asked to participate in the virtual intervention, consisting of six-weekly group classes via Zoom, and six-weekly personalized teleconsultations (via phone call or Zoom) at a suitable time for both participants and CHWs. Study participants will receive 6 linguistically and ethnically concordant weekly two-hour group classes and personalized teleconsultations led by CHWs. The total time commitment for Group 2 will be a maximum of 20 hours (6 two-hour group classes, + 6 one hour personal session, + 2 half hour phone calls), over the next 6 weeks.
  Interventions: Behavioral: Community Health Worker led curriculum

INTERVENTIONS:
Behavioral: Community Health Worker led curriculum — The intervention arm will consist of a CHW-based health educational program via Zoom, where participants will be provided with information about COVID-19, COVID-19 resources and services in Los Angeles County, and engagement with Los Angeles County Department of Health Services CHWs who will lead the curriculum and be available to answer questions of the intervention arm patients.
  Arms: Intervention Arm - CHW-led curriculum (Group 2)

SUMMARY:
The objective of this study is to compare the results of a COVID-19 specific curriculum led by LACDHS Community Health Workers (CHWs) from these same communities of safety-net patients to effectively increase COVID-19 testing and vaccination for individual patients, and to facilitate needed healthcare in a timely manner for the safety net health system, and to develop a sustained public health presence in these communities to build trust and preparedness for critical COVID-19 related future needs.

DETAILED DESCRIPTION:
This study represents the third aim of a grant with three aims. The study used unsupervised machine learning and qualitative interviews to develop a CHW intervention for this aim. The aim will compare and evaluate a Community Health Worker-led curriculum aimed to identify and address barriers to COVID-19 testing and vaccination among LACDHS safety-net patients.

For the study, the investigators will recruit 66 eligible safety-net patients for a COVID-19 specific curriculum, provided by Community Health Workers at Los Angeles County Department of Health Services. The study will take place remotely over the course of 6-weeks. Utilizing a randomized control design among African American and Latinx safety net patients, will assess the effect of the CHW hypothesis-driven intervention on trust, self-efficacy, and intent to participate in COVID-19 testing and vaccination.

The remote CHW intervention that the study participants will participate in and be compensated for is a pilot program intended to provide additional CHW training. Monthly calls from LACDHS to remind them of COVID-19 vaccination are standard of care for all empaneled LACDHS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years and older
* Self-identify as African American or Latinx
* English Speaking
* Receives primary or specialty care treatment at an LACDHS facility
* Has either not completed lab orders for COVID-19 testing and/or vaccination at an LACDHS facility
* Have reliable internet access

Exclusion Criteria:

* Not meeting the inclusion criteria listed above

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Project Survey: Phenx toolkit - Worry about COVID | Six weeks from start of project
  In a 4-point Likert scale, we will ask questions about their worry and concern about getting infected with COVID from "extremely concerned, somewhat concerned, neutral, not concerned" Measure three key measures: trust, self-efficacy, and intent to participate in COVID-19 testing and vaccination. Consolidated pre- and post- surveys (Name: Project Survey) will measure participants' intentions of getting vaccinated and tested for COVID-19.
Project Survey: Phenx toolkit - Attitudes and Behavior | Six weeks from start of project
  In a 5 point Likert scale, questions will ask about attitudes, and behaviors regarding COVID, from "very likely, somewhat likely, neutral, somewhat unlikely, and very unlikely" Measure three key measures: trust, self-efficacy, and intent to participate in COVID-19 testing and vaccination. Consolidated pre- and post- surveys (Name: Project Survey) will measure participants' intentions of getting vaccinated and tested for COVID-19.
Project Survey: Phenx toolkit - Perceived Coronavirus Threat | Six weeks from start of project
  In a 4-point Likert scale, we will ask questions about their perceived Coronavirus threat "extremely concerned, somewhat concerned, neutral, not concerned" Measure three key measures: trust, self-efficacy, and intent to participate in COVID-19 testing and vaccination. Consolidated pre- and post- surveys (Name: Project Survey) will measure participants' intentions of getting vaccinated and tested for COVID-19.

SECONDARY OUTCOMES:
Project Survey: Phenx toolkit - Intent to participate in COVID testing and vaccination | Six weeks from start of project
  assessed by a single declarative item using a four-point scale (very likely, somewhat likely, somewhat not likely, very not likely). Consolidated pre- and post- surveys (Name: Project Survey) will measure participants' intentions of getting vaccinated and tested for COVID-19.
Pre and Post Program Survey: Medical Mistrust Scale | Six weeks from start of project
  Trust will be measured using 8 adapted items from the Medical Mistrust scale, with a list of statements asking about general feelins about the healthcare systems, answers will be "strongly disagree, disagree, neutral, agree, strongly agree"
Sherer, et al.'s General Self-Efficacy Scale | Six weeks from start of project
  It contains 17 items that are rated on a 5-point Likert-type scale ranging from agree strongly to disagree strongly and are intended to assess a "general set of expectations that the individual carries into new situations"

CONTACTS AND LOCATIONS:
Overall Officials: Sheba George, PhD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (2):
- United States (2):
  - Los Angeles Department of Public Health, Los Angeles, California
  - Charles Drew University of Medicine and Science, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
The study falls is managed through the RADxUP program and such it is required for supplement grant projects to share their data dictionaries to the RADx Data Hub.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available at the end of study and will be uploaded to the RADxUP Data Hub, managed by Duke Coordinating Center
Access Criteria: Only authorized RADxUP personnel will be able to access the IPD. The link below details how the COVID RADx Data Hub is a centralized, secure repository to store, search for and interrogate vast amounts of de-identified data related to COVID-19 testing and vaccination.
URL: https://radx-up.org/research/cdes/

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT05473936/Prot_000.pdf
  • Informed Consent Form (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT05473936/ICF_001.pdf